CLINICAL TRIAL: NCT00301158
Title: Involving Adolescents in Physical Activity Promotion
Brief Title: Promoting Physical Activity In After-School Programs for Urban Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Montclair State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Prevention
Other Study IDs: CDR0000455588; MSUHNS-0003669; FWA00005270
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Counseling; Early Intervention, Educational

INTERVENTIONS:
Behavioral: exercise intervention
Other: counseling intervention
Other: educational intervention
Procedure: complementary or alternative medicine procedure

SUMMARY:
RATIONALE: Physical activity may lower the risk of some types of cancer and other chronic diseases.

PURPOSE: This clinical trial is studying ways to increase physical activity in urban adolescents who attend after-school programs.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Develop educational, promotional, and evaluation materials for use in promoting physical activity (PA) in community-based after-school programs by multiethnic, urban adolescents.
* Develop a series of workshops for promoting physical activities (PAs) that are "a good fit" in after-school programs for these participants.
* Determine a small set of feasibility tests as a first step towards pursuing funding for a full-scale experimental study.
* Development of print materials for a series of skills-building workshops for these participants.
* Development of evaluation materials, including self-report survey questions and structured interview protocols for qualitative assessment of participants' skills in identifying PAs that are a "good fit" for them.

OUTLINE: Youth participants will be assigned to one of two groups and may be involved in one or more research activities conducted during after-school hours at a community-based, after-school program site.

* Focus group: Participants, consisting of 5-8 adolescents per focus group, either all male or all female, attend a single audiotaped focus group with a trained moderator for 60 minutes. Participants complete an anonymous participant information form, and explore their perceptions of physical activity (PA), perceptions of audience segments among peers that would be appropriate for tailoring physical promotions, and responses to images and graphic designs for use in developing print materials. Some participants may also be eligible to participate in a second focus group and the survey if interested.
* One-on-one interview: Participants attend a one-on-one audiotaped individual interview with a trained interviewer for 60 minutes. Participants in the first set of interviews explore their perceptions of PA, their perceptions of the concept of finding PAs that are "a good fit", and their perceptions of audience segmentation for promoting PA. In the second set of interviews, participants test a protocol for qualitative assessment of adolescents' skills in assessing "good fit" of PA. Participants are involved in a series of visual and written scenarios depicting a variety of PAs, and use a structured interview format to identify the PA they most or least enjoy. Participants will also be asked to elaborate on criteria and experiences on which they based their decisions. Participants may also participate in the survey if interested.
* Survey: Participants complete a paper and pencil 60-minute questionnaire about PA behaviors, attitudes, environments, and person-physical activity skills (i.e., skills in finding PAs that are "a good fit"). Two weeks later, participants are asked to complete a second questionnaire.
* Key informant interview (adult): Participants attend a 60-minute, audiotaped interview with a trained interviewer that focuses on respondents' perceptions of the PA-related attitudes, behaviors, strengths, and barriers of the young adolescents who participate in their program, the respondents' experiences with promoting PA in their program participants, and respondents' suggestions for program elements and logistics to enhance the feasibility and effectiveness of after-school workshops to promote PA.
* Workshop pilot testing: After data collection from the above field work is completed, 1-2 workshop activities are conducted in cooperation with program leaders at community-based, after-school programs.

PROJECTED ACCRUAL: Approximately 420 participants (400 adolescents and 20 adults) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Noninstitutionalized, community-residing youth living in and attending after-school programs in New York City or Newark, NJ OR
* After-school program leaders at community agencies (i.e., adults) who participate in key informant interviews

PATIENT CHARACTERISTICS:

* Any racial or ethnic background

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 420 (Estimated)
Dates: Start 2004-09; Primary Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Behavior changes regarding physical activity by self-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Amanda S. Birnbaum, PhD, MPH, Study Chair — Montclair State University
Locations (1):
- Health and Nutrition Sciences at Montclair State University, Montclair, New Jersey, United States